CLINICAL TRIAL: NCT05085379
Title: Optical Coherence Tomography of the Middle Ear Using Ossiview
Status: Withdrawn | Type: Observational
Why Stopped: No Subjects enrolled
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Other Study IDs: 262886.
Record Dates: First submitted 2021-10-07; First posted 2021-10-20 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2023-03

CONDITIONS: Middle Ear Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: Ossiview — Imaging of the ear using Optical Coherence Tomography

SUMMARY:
The aim of this study is to understand the diagnostic applications for this imaging technology and identify particular disorders to target for future clinical investigations. Images obtained with the Ossiview device will be correlated to other standard of care (SoC) testing including microscopic otoscopy, CT scans, MRIs, audiologic testing results, and surgical and pathology reports.

DETAILED DESCRIPTION:
Optical Coherence Tomography (OCT) is an optical imaging technique that uses a low-coherence interferometer to produce depth-resolved scans in tissue. This study will explore the utility of this technology in otology patients presenting with various pathologies as well as normal subjects.

ELIGIBILITY:
Inclusion Criteria

* Age ≥18 years
* Ability to understand the consent process with adequate language and cognitive communication ability
* Presence of one of the pathologies (either currently or in the past) above or healthy control

Exclusion Criteria

* Narrow or stenotic external meatus (ear canal)
* Movement disorder causing inability to keep head still during imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Target pathologies in the subject population are subjects with:
  * Chronic ear disease
  * Suspected mixed hearing loss or sensorineural hearing loss
  * Otosclerosis
  * Suspected or confirmed conductive hearing loss
  * Cholesteatoma
  * Otitis Media
  * Ossicular erosion
  * Perforated TM
  * Ossicular fixation
  * Functioning middle ear prosthesis
  * Failed middle ear prosthesis
  * Head/Ear trauma patients
  * Cochlear implant patients
  * Previous tympanoplasty
  * Vascular defects
  * Tympanosclerosis
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-11-02 (Actual); Primary Completion 2023-11-02 (Actual); Study Completion 2023-11-02 (Actual)

PRIMARY OUTCOMES:
Diagnostic correlation with microscopic otoscopy | 6 months
  Comparison of Diagnostic ability to other standard of care (SoC) testing - microscopic otoscopy
Diagnostic correlation with CT scans | 6 months
  Comparison of Diagnostic ability to other standard of care (SoC) testing - CT scans
Diagnostic correlation with Magnetic Resonance Imaging (MRI)s | 6 months
  Comparison of Diagnostic ability to other standard of care (SoC) testing - MRIs
Diagnostic correlation with audiologic testing results | 6 months
  Comparison of Diagnostic ability to other standard of care (SoC) testing - audiologic testing results
Diagnostic correlation with surgical reports | 6 months
  Comparison of Diagnostic ability to other standard of care (SoC) testing - surgical reports
Diagnostic correlation with pathology reports | 6 months
  Comparison of Diagnostic ability to other standard of care (SoC) testing - pathology reports

CONTACTS AND LOCATIONS:
Overall Officials: Deanne King, MD, PhD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, AR, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No